CLINICAL TRIAL: NCT02247206
Title: Voice Over Internet Protocol Delivered Behavior Therapy for Tourette Syndrome
Brief Title: VoIP Delivered Behavior Therapy for Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Emily Ricketts, Doctoral Student, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIL105611; F31MH096375-01 (NIH); 5F31MH096375-02 (NIH)
Record Dates: First submitted 2014-09-15; First posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Tourette Syndrome; Chronic Tic Disorder
Keywords: Tourette Syndrome; tic disorders; behavior therapy; web-based videoconferencing; VoIP
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavior Therapy for Tics (CBIT) (Experimental): The child 1) learns to become more aware of any sensations, or urges that may trigger tics, and 2) learn some other behavior (competing response) to do every time he/she feels the urge to tic. The child's parent is trained to provide prompts and praise for use of the competing response. The parent and family also receive psychoeducation about tics, and learn ways to reduce the impact of environmental stimuli on tic severity. The child learns relaxation techniques to reduce stress and make it easier for him/her to resist his or her tics. Prior to treatment sessions, the parent and child spend about 10 minutes discussing with the therapist any problematic issues he/she is having. At the end of treatment sessions the child is assigned some tasks to practice prior to the next session.
  Interventions: Behavioral: Behavior Therapy for Tics (CBIT)
- Waitlist-control Group (No Intervention): Participants in the waitlist-control group, do not receive behavior therapy for tics or any other treatment during the 10-week acute treatment period. Instead they child are placed on a waitlist to receive videoconference-delivered treatment following the end of the study period.

INTERVENTIONS:
Behavioral: Behavior Therapy for Tics (CBIT) — CBIT is an 8-session 10-week behavioral treatment for chronic tic disorders, including Tourette Syndrome. The first two sessions are 90 minutes, with subsequent sessions lasting 60 minutes. The treatment consists of Habit Reversal Training (awareness training, competing response training, and social support), and function-based assessment to reduce the impact of environmental or other stimuli on tic severity. The treatment also consists of relaxation techniques to reduce tic-related stress and tension, and behavioral rewards to motivate treatment compliance.
  Other Names: Comprehensive Behavioral Intervention for Tics (CBIT); Habit Reversal Training (HRT)
  Arms: Behavior Therapy for Tics (CBIT)

SUMMARY:
The purpose of this research is to examine the preliminary efficacy, feasibility, and acceptability of Voice over Internet Protocol delivered behavior therapy for Tourette Syndrome through in a randomized waitlist-controlled trial.

DETAILED DESCRIPTION:
A Comprehensive Behavioral Intervention for Tics (CBIT) is an emerging treatment for children with Tourette Syndrome (TS) and has been shown to be efficacious in separate randomized trials with children and adults; however, many families of children with TS are prevented from accessing it due to limited availability of adequately trained treatment providers. Recent research has shown that videoconference-delivered CBIT is as effective as face to face delivery, and that both modalities are efficacious. Despite its effectiveness, traditional videoconferencing has limitations including lack of portability, ease of access, the need for third party clinics, and cost. A newer, more convenient alternative to increase access is the use of Voice over Internet Protocol (VoIP) transmission, allowing for the direct delivery of CBIT to patients' homes.

Therefore the objective of this study (the final phase of a three-phase project) is to establish the preliminary efficacy of VoIP-modified CBIT for reducing tics in children with TS relative to a waitlist-control. Twenty children (ages 9-17) with TS or Chronic Tic Disorder as a primary diagnosis will be recruited for a randomized, observer-blind, waitlist controlled trial of VoIP-delivered CBIT. Participants will be randomly assigned to 8 weekly sessions of CBIT-VoIP over a 10-week acute treatment period, or waitlist control condition. As an exploratory aim, the current study will investigate potential correlates of treatment outcome, including home computer equipment available (i.e., web camera type, microphone type, internet upload speed, and type of internet connection), prior computer experience, and comfort with study computer equipment.

ELIGIBILITY:
Inclusion Criteria:

* Resides in the state of Wisconsin
* Ages 8-17
* Meets DSM-IV-TR diagnostic criteria for Chronic Tic Disorder (CMVT or TS)
* Clinical global Impressions - Severity Score greater than or equal to 4 (moderately ill)
* YGTSS Total Score greater than or equal to 14 and less than 30 OR Total Score greater than or equal to 10 and less than 20 if CTD with motor tics only
* Unmedicated or on stable medication treatment for tics, OCD, ADHD, anxiety, and/or depressive disorder for at least 6 weeks, with no planned changes for duration of study participation
* Fluent English speaker

Exclusion Criteria:

* YGTSS Total Tic Score > 30 (for any score exceeding 30 on the YGTSS, the research team determined the appropriateness of the patient's participation in the study, taking into account the patient's global functioning)
* WASI-Vocab subtest T-Score < 37
* DSM-IV substance abuse or dependence or Conduct Disorder within the past 3 months
* Lifetime DSM-IV diagnosis of Pervasive developmental disorder, Mania, or Psychotic Disorder
* Any serious psychiatric, psychosocial, or neurological condition requiring immediate treatment other than that provided in the current
* Previous treatment with HRT for tics (four or more sessions)
* Lack of a functional, and accessible home computer, and high speed (i.e., cable/DSL) internet connection
* Refusal to sign a release of information form for the child's local primary care physician, mental health professional, or neurologist.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Yale Global Tic Severity Scale (YGTSS) total tic severity scores at 10 weeks | Baseline, 10-week (post-treatment)
  The YGTSS is a clinician-rated tic severity measure, featuring a total severity score, with a rating from 0 to 50, and independent subtotals for motor and vocal tics each with ratings from 0 to 25. It also features a tic-related 0-50 point impairment scale.

SECONDARY OUTCOMES:
Change from baseline on the Clinical Global Impressions-Severity scale at 10 weeks | Baseline, 10-week (post-treatment)
  The CGI-S is a clinician-rated measure of patient global impairment.
Treatment response rate using the Clinical Global Impressions-Improvement scale at 10 weeks | 10-week (post-treatment)
  The CGI-I is a rating of patient improvement compared to baseline. Scores of Much (2) or Very Much (1) Improved indicate positive treatment response in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Ricketts, PhD, Principal Investigator — University of Wisconsin, Milwaukee; Douglas W Woods, PhD, Study Director — Texas A&M University; Michael B Himle, PhD, Study Chair — University of Utah
Locations (1):
- University of Wisconsin-Milwaukee Psychology Department, Milwaukee, Wisconsin, United States